CLINICAL TRIAL: NCT05210985
Title: Examination of the Relationship Between Home Affordances With Motor Development and Sensory Processing in Preterm Infants
Brief Title: Examination of the Relationship Between Home Affordances With Development
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia Eraslan, principal investigator, Gazi University
Other Study IDs: Home affordances
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Preterm Birth
Keywords: Preterm; home affordances; Sensory development; motor development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — motor and sensory development assesment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premature babies: Fifty infants between 4-18 months with a history of premature birth and with the consent of their parents will be included in the study. Babies with the chromosomal anomalies, serious congenital problems, and whose parents are not willing to work will not be included in the study.
  Interventions: Behavioral: Affordances in the Home Environment for Motor Development-Infant Scale; Behavioral: Peabody Developmental Motor Scales-2; Behavioral: Test Of Sensory Functions In Infants (Tsfı)

INTERVENTIONS:
Behavioral: Affordances in the Home Environment for Motor Development-Infant Scale — Affordances in the Home Environment for Motor Development-Infant Scale is a parent-filled assessment to determine the nature and amount of factors affecting infant motor skill development in the home environment, including the availability of toys, materials, and the availability of spaces.
Behavioral: Peabody Developmental Motor Scales-2 — Peabody Developmental Motor Scales | Second Edition (PDMS-2) combines in-depth assessment with training or remediation of gross and fine motor skills of children from birth through 5 years.
Behavioral: Test Of Sensory Functions In Infants (Tsfı) — This test helps you identify infants with sensory integrative dysfunction-including those at risk for developing learning disabilities as they grow older. The TSFI provides objective criteria that allow you to determine whether, and to what extent, an infant has deficits in sensory functioning. Designed for use with children from 4 months to 18 months old, the TSFI provides an overall measure of sensory processing and reactivity, as well as scores on the following subdomains: Reactivity to Tactile Deep Pressure Visual Tactile Integration Adaptive Motor Function Ocular Motor Control Reactivity to Vestibular Stimulation

SUMMARY:
Babies with a history of premature birth and low birth weight are at risk for developmental disorders. These infants may have motor, cognitive and behavioral problems compared to their term peers. Although advances in technology lead to an increase in survival rate, 50% of these infants may have developmental delays in motor, cognitive and behavioral areas. Premature birth does not accelerate any of the early sensory development processes, but exposure to intense, unusual stimuli of unusual character may delay or inhibit sensory development. Therefore, children born prematurely may be at risk in terms of sensory processing. The physical, sensory and social environment of the infant and young child is critical in supporting the healthy and appropriate development of the brain and nerve-sensory systems.

DETAILED DESCRIPTION:
A newborn baby reacts involuntarily or reflexively to its environment. During the first few years of life, through physical growth and learning experiences, the child learns to participate actively in the world. Motor skills and sensory experiences begin to develop after birth, and development continues as children grow. Having good motor control also helps children explore the world around them, which can help many other areas of development. There are many environmental and biological factors that affect motor development. Especially the home environment where the child spends most of his time is one of the key factors affecting motor development. The home environment is known to be a very important factor for motor development in infants. At the same time, the variety of equipment and environmental conditions help children provide different sensory experiences. Exploring the home environment can have important developmental implications, as it is common practice for physiotherapists to advise patients on home activities. Environmental factors can affect the motor development of preterm children as well as other developmental areas. The number of studies examining the effects of environmental factors on motor and sensory development in preterm infants is limited in the literature. This study was planned to examine whether there is a relationship between the environmental conditions and equipment variety and the motor and sensory development of the preterm child.

ELIGIBILITY:
Inclusion Criteria: Fifty infants between 4-18 months with a history of premature birth and with the consent of their parents will be included in the study.

Exclusion Criteria:

Babies with chromosomal anomaly, serious congenital problems and whose parents are not willing to work will not be included in the study.

Ages: 4 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: It was planned to include infants who applied to Gazi University Faculty of Health Sciences Physiotherapy and Rehabilitation Department Pediatric Rehabilitation unit in the study. Fifty infants between 4-18 months with a history of premature birth and with the consent of their parents will be included in the study. Babies with chromosomal anomalies, serious congenital problems, and whose parents are not willing to work will not be included in the study. In the evaluations, the demographic characteristics of the babies (sex, gestational age, corrected age, birth weight, parental information, mother's pregnancy type, pregnancy history, Apgar score, treatments received, history of staying in the intensive care unit, risk factors) will be recorded in the file and by interviewing the family.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Affordances in the Home Environment for Motor Development-Infant Scale | 4-18 months
  Affordances in the Home Environment for Motor Development-Infant Scale is a parent-filled assessment to determine the nature and amount of factors affecting infant motor skill development in the home environment, including the availability of toys, materials, and the availability of spaces. The scale consists of 41 items in total. For babies aged 3-12 months, questions up to the first 32 items are answered. It is stated that other substances are not suitable for babies under 12 months. All substances are applied to babies between 12-18 months. Questions answered as yes or no are scored as 0.1 (0: no, 1: yes). Other questions are scored as 0, 1, 2, 3. For babies up to 12 months, a total of 66 points is obtained. For babies older than 12 months, a total of 93 points is obtained. A higher score indicates better environmental enrichment.
Test of Sensory Functıons ın Infants | 4-18 months
  This test helps you identify infants with sensory integrative dysfunction-including those at risk for developing learning disabilities as they grow older. All subtests consist of a total of 24 items. In the tactile deep pressure response section, it is scored as 0: reverse response, 1: mild defensive response, and 2: integrated response. In the adaptive motor response section, it is scored as 0: no response, 1: disorganized, 2: partial, 3: organized. In the visual-tactile integration section, it is scored as 0: hyperactive, 1: hyporeactive, and 2: normal. The oculomotor test section is scored as 0: no response or poorly integrated, 1: well integrated. Response to vestibular stimulation is scored as 0: adverse response, 1: mild defensive response, and 2: integrated response. The total score ranges from 0 to 49. In 10-12-month-old babies, 44-49 points indicate good sensory function, 41-43 points indicate risky status, 0-40 points sensory processing problem.
Peabody Developmental Motor Scales | Second Edition | 4-18 months
  Peabody Developmental Motor Scales | Second Edition (PDMS-2) combines in-depth assessment with training or remediation of gross and fine motor skills of children from birth through 5 years. It consists of gross motor and fine motor parts. The Gross motor section includes 151 items from 4 subtests: reflexes, stasis, locomotion, and object manipulation. The fine motor section consists of 2 subtests and 98 items: comprehension and visual-motor integration. The total motor part is the sum of the items in the gross and fine 25 motor parts. Items are scored with 0, 1, and 2 points. When the child performs the item according to the specified item criteria, 2 points are given. 1 point is awarded when the behavior occurs but the criteria for successful performance are not fully met. A score of 0 is given when the child is unable to try the item or does not reveal any skills when he tries it. Results are expressed as a raw score, standard score, or total motor score.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Eraslan, Principal Investigator — Gazi University
Locations (1):
- Rabia Eraslan, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodward LJ, Anderson PJ, Austin NC, Howard K, Inder TE. Neonatal MRI to predict neurodevelopmental outcomes in preterm infants. N Engl J Med. 2006 Aug 17;355(7):685-94. doi: 10.1056/NEJMoa053792. PMID 16914704
- [Background] Noble Y, Boyd R. Neonatal assessments for the preterm infant up to 4 months corrected age: a systematic review. Dev Med Child Neurol. 2012 Feb;54(2):129-39. doi: 10.1111/j.1469-8749.2010.03903.x. Epub 2011 Dec 5. PMID 22142216
- [Background] Kaya-Kara O, Kerem-Gunel M, Yigit S. Correlation of the Bayley scales of infant-toddler development-3rd edition and neuro-sensory motor assessment in preterm infants during the first year of life. Turk J Pediatr. 2019;61(3):399-406. doi: 10.24953/turkjped.2019.03.012. PMID 31916718
- [Background] Cacola PM, Gabbard C, Montebelo MI, Santos DC. Further Development and Validation of the Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS). Phys Ther. 2015 Jun;95(6):901-23. doi: 10.2522/ptj.20140011. Epub 2014 Dec 18. PMID 25524875
- [Background] Cacola P, Gabbard C, Santos DC, Batistela AC. Development of the Affordances in the Home Environment for Motor Development-Infant Scale. Pediatr Int. 2011 Dec;53(6):820-5. doi: 10.1111/j.1442-200X.2011.03386.x. PMID 21507146